CLINICAL TRIAL: NCT01357499
Title: Effects of Lower Leg Remote Ischemic Preconditioning in Combination With Electric Muscle Stimulation in Elective Coronary Artery Revascularisation
Brief Title: Lower Leg Remote Ischemic Preconditioning in Elective Percutaneous Coronary Intervention (PCI)
Acronym: REMOTE
Status: Withdrawn | Type: Observational
Why Stopped: PI left center
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Marcus Doerr, MD, University Medicine Greifswald
Other Study IDs: 1-reinthaler
Record Dates: First submitted 2011-05-10; First posted 2011-05-20 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood samples (10 ml) will be taken from the femoral vein of the preconditioned leg immediately before and after the preconditioning cycles.
  Also arterial blood samples (10 ml)will be taken immediately before and after the preconditioning cycle.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- control group: A Blood pressure cuff and and the muscle stimulator pads will be applied to one lower leg but without inflating the cuff and without stimulating the muscle. Now 25 minutes will have to pass by before beginning the coronary angioplasty.
- intervention group 1: A Blood pressure cuff and and the muscle stimulator pads will be applied to one lower leg. The blood pressure Cuff will be inflated with 200 mmHg for 5 minutes. Next reperfusion will be allowed for 5 minutes. This cycle will be repeated for 3 times. There will be no electrical muscle stimulation in this group.
  Interventions: Device: blood pressure cuff
- intervention group 2: A Blood pressure cuff and the muscle stimulator pads will be applied to one lower leg. The blood pressure Cuff will be inflated with 200 mmHg for 5 minutes. Next reperfusion will be allowed for 5 minutes. This cycle will be repeated for 3 times. In addition electrical muscle stimulation will be performed throughout the whole preconditioning cycle
  Interventions: Device: blood pressure cuff + electric muscle stimulator

INTERVENTIONS:
Device: blood pressure cuff — A Blood pressure cuff and and the muscle stimulator pads will be applied to one lower leg. The blood pressure cuff will be inflated with 200 mmHg for 5 minutes. Next reperfusion will be allowed for 5 minutes. This cycle will be repeated for 3 times.
  Groups: intervention group 1
Device: blood pressure cuff + electric muscle stimulator — A Blood pressure cuff and and the muscle stimulator pads will be applied to one lower leg. The blood pressure Cuff will be inflated with 200 mmHg for 5 minutes. Next reperfusion will be allowed for 5 minutes. This cycle will be repeated for 3 times. In addition electrical muscle stimulation will be performed throughout the whole preconditioning cycle.
  Groups: intervention group 2

SUMMARY:
The purpose of this study is to investigate if remote ischemic preconditioning by combining limb ischaemia with electric muscle stimulation of the ischemic muscle provokes better results in preconditioning the human heart than limb ischaemia alone does.

DETAILED DESCRIPTION:
It has been demonstrated that protection from ischemia reperfusion can be achieved by brief periods of ischemia applied at a remote site during an injurious ischemic event (remote postconditioning). The purpose of this study is to investigate if the combination of brief periods of limb ischemia in combination with electric muscle stimulation at the same site could exceed the preconditioning effect of limb ischemia alone.

Therefore the investigators thought to perform 2 different forms of remote ischaemic preconditioning in patients undergoing elective coronary angioplasty.

In the first patient group a blood pressure cuff will be applied at the lower leg. Ischemia will be induced by inflating the cuff to a pressure of 200 mmHg for 5 minutes. Afterwards reperfusion will be allowed for further 5 minutes. This cycle will be repeated 3 times.

In a second patient group electric muscle stimulation at the same site (HiToP 191) will be performed additionally throughout the whole preconditioning cycle.

After preconditioning, the percutaneous coronary intervention (PCI) will be performed by 3 PCI-ballon inflations, each lasting for 2 minutes. Between the inflations coronary reperfusion will be allowed for 5 minutes.

The Effects of preconditioning will be evaluated by analysing the ST-deviation, caused by angioplasty in an intracoronary (derived by PCI wire) and surface ecg.

Also the maximum of chest pain during the 3 inflation cycles and troponin levels 24 h after PCI will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* planned PCI of one of the main coronary artery (artery diameter distal of the stenotic area at least 2,5 mm)
* patient age 18 years or older
* stable angina pectoris symptoms

Exclusion Criteria:

* presence of collateral vessels
* electrocardiographic bundle branch blocks
* multiple coronary stenosis
* occlusion of a coronary artery
* renal insufficiency (GFR (MDRD) < 50 ml/min/1,73 m2)
* presence of coronary bypass grafts
* history or presence of myocardial infarction.
* echocardiographic signs of left ventricular hypertrophy (septal and/or posterior wall diameter greater than 14 mm)
* some sort of medications (adenosine, morphine and derivates, immunosuppressive agents, oral antibiotics, theophyllin, alpha receptor blockers)
* peripheral arterial disease
* exercise tests performed within 24 h before study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective PCI fulfilling the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
ST deviation | 120 seconds after angioplasty
  Immediately after the preconditioning cycle the PCI ballon will be positioned in the coronary artery lesion and inflated for 2 minutes followed by 5 minutes of reperfusion. This cycle will be repeated for 3 times without any interruption. Intracoronary ECGs and 12 lead surface ecgs will be taken immediately before and at the end of each ballon inflation (two minutes after beginning the intracoronary ballon inflation). after taking the ecgs the ballon will be deflated.
  The st-deviations will be analysed.

SECONDARY OUTCOMES:
troponin I | 24 hours after PCI
  Troponin levels will be evaluated 24 h after PCI
chest pain (Maximum) | time period 2 minutes
  the maximal chest pain occuring during each of the Pci balloon inflations will be documented as a number out of 10. 0 is determined as no pain and 10 is determined as the heaviest pain which the patient ever experienced. A specific timepoint has not been defined.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Reinthaler, MD, Principal Investigator — Ernst Moritz Arndt University Greifswald; Thorsten Reffelmann, MD, Principal Investigator — Ernst Moritz Arndt University Greifswald
Locations (1):
- Ernst Moritz Arndt Universität Greifswald, Greifswald, MVP, Germany